CLINICAL TRIAL: NCT00795561
Title: Randomized Controlled Trial of Day Care Versus Inpatient Management of Nausea and Vomiting of Pregnancy
Brief Title: Management of Nausea and Vomiting of Pregnancy
Acronym: DIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Fergus McCarthy, Research Fellow, Specialist Registrar Obstetrics and Gynaecology, University College Cork
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISRCTN05023126; ISRCTN05023126
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Hyperemesis Gravidarum; Nausea; Vomiting; Pregnancy
Keywords: Hyperemesis gravidarum; nausea; vomiting; pregnancy; day care; inpatient management; Nausea and vomiting of pregnancy
MeSH Terms: conditions — Hyperemesis Gravidarum; Nausea; Vomiting | interventions — Day Care, Medical; Inosine Monophosphate; Patient Admission

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Day care (Experimental): Patients randomised to day care treatment of NVP will be instructed to present to the day services unit where they will receive a pre-agreed fluid and anti emetic regimen.
  Interventions: Procedure: Day care
- Inpatient (Active Comparator): Patients randomised to inpatient management of NVP will be admitted to hospital where they will receive a pre-agreed fluid and anti emetic regimen.
  Interventions: Procedure: Inpatient

INTERVENTIONS:
Procedure: Day care — Patients randomised to day care treatment of NVP will be instructed to present to the day services unit where they will receive a pre-agreed fluid and anti emetic regimen.
  Other Names: day unit; day services
  Arms: Day care
Procedure: Inpatient — Patients randomised to inpatient management of NVP will be admitted to hospital where they will receive a pre-agreed fluid and anti emetic regimen.
  Other Names: admission
  Arms: Inpatient

SUMMARY:
Upto 80% of all pregnant women experience some form of nausea and vomiting (NVP) during their pregnancy. Hyperemesis gravidarum, a more severe form of NVP affects approximately 0.3- 2.0% of pregnancies and is the commonest indication for admission to hospital in the first half of pregnancy and second only to preterm labor as a cause of hospitalization overall. According to the Hyperemesis Education and Research Foundation, conservative estimates indicate that HG can cost a minimum of $200 million annually in house hospitalizations in the United States of America. The investigators aim to conduct a randomized controlled trial to test the hypothesis that the availability of day care services for the initial treatment of NVP reduces the mean duration of stay in hospital by 1 day and results in significantly greater patient satisfaction compared with standard inpatient management.

DETAILED DESCRIPTION:
Upto 80% of all pregnant women experience some form of nausea and vomiting during their pregnancy (NVP). The International Statistical Classification of Disease and Related Health Problems ICD-10 defines hyperemesis gravidarum (HG) as persistent and excessive vomiting starting before the end of the 22nd week of gestation, and further subdivides the condition into mild and severe, severe being associated with metabolic disturbances such as carbohydrate depletion, dehydration or electrolyte imbalance. HG is a diagnosis of exclusion, characterized by prolonged and severe nausea and vomiting, dehydration, large ketonuria and > 5% bodyweight loss.

HG affects approximately 0.3- 2.0% of pregnancies and is the commonest indication for admission to hospital in the first half of pregnancy and second only to preterm labor as a cause of hospitalisation overall. According to the Hyperemesis Education and Research Foundation, conservative estimates indicate that HG can cost a minimum of $200 million annually in house hospitalizations in the United states. Taking into account other factors such as emergency room treatments, potential complications of severe HG and the fact that up to 35% of women with paid employment will lose time from work through nausea the actual cost of NVP to the economy is significantly higher.

NVP can be extremely debilitating for the patient and if inadequately managed can cause significant morbidities including malnutrition and electrolyte imbalances, thrombosis, Wernicke's encephalopathy, depressive illness and poor pregnancy outcomes such as prematurity and small for gestational age fetuses.

Day care has proven to be beneficial and safe mode of care for patients in other clinical settings. Studies have demonstrated that day care management of patients with NVP appears acceptable and feasible but no systematic reviews or randomized controlled trials have been performed which examine the effects of introducing day care on rates of hospital admission, duration of inpatient stay and patient satisfaction.

We aim to conduct a prospective open label randomized controlled trial to test the hypothesis that the availability of day care services for the initial treatment of NVP reduces the mean duration of stay in hospital by 1 day (28.6%) and results in significantly greater patient satisfaction compared with standard inpatient management.

The null hypothesis states there is no difference in the amount of inpatient hospital days when women with NVP are treated initially in day care or by standard inpatient admission.

All pregnant women under 22 weeks gestation, who have not already been treated for NVP in their current pregnancy, presenting with the diagnosis of NVP are eligible for inclusion in the trial. The treatment group will be day care treatment of NVP. The comparison group will be the inpatient treatment of NVP.

ELIGIBILITY:
Inclusion Criteria:

Women (no age limits) will be admitted to the study if they have two or more of the following criteria

* Ongoing viable intrauterine pregnancy/ pregnancies < 22 weeks gestation
* Persistent vomiting (>x3 episodes/ 24 hours) not attributable to other causes
* Severe nausea not attributable to other causes.
* Dehydration diagnosed by the presence of ketonuria.
* Electrolyte imbalance not attributable to other causes.

Exclusion Criteria:

Women will not be admitted to the study if any of the following criteria are present.

* Women with a confirmed urinary tract infection (mid stream urine isolation of a single strain of uropathogen >105 bacteria/ml)
* Women with molar pregnancies
* Women with non viable pregnancies.
* Women who have already received treatment for NVP outside of this trial.
* Pregnant women who present who will not be booking at CUMH for their pregnancy or are not resident in the South West of Ireland i.e. day care treatment is not an option.
* Women who do not have a good understanding of English.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the number of inpatient nights spent in hospital secondary to NVP from initial presentation until 22 weeks gestation. An inpatient night will be defined as requiring an inpatient bed between the hours of 20.00 and 08.00. | Following discharge

SECONDARY OUTCOMES:
Total number of hours spent in hospital secondary to NVP from initial presentation until 22 weeks gestation. | 22 weeks gestation
Total amount of intravenous fluids administered secondary to NVP from initial presentation until 22 weeks gestation | 22 weeks gestation
Total amount of anti-emetics administered secondary to NVP from initial presentation until 22 weeks gestation. | 22 weeks gestation
Total Multivitamin complexes administered secondary to NVP from initial presentation until 22 weeks gestation | 22 weeks gestation
Patient satisfaction will be measured by the Client Satisfaction Questionnaire. | Following first presentation
Incidence of miscarriage | 22 weeks gestation
Infant birth weight at delivery | Following delivery
Gestational age at delivery. | following delivery
Total days lost at work secondary to NVP from initial presentation until 22 weeks gestation. (Asked at 16 weeks gestation) | 16 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: John R Higgins, MD, Principal Investigator — Cork University Maternity Hospital
Locations (1):
- Department of Obstetrics and Gynaecology, Cork University Maternity Hospital, Cork, Ireland

REFERENCES:
- [Background] Gazmararian JA, Petersen R, Jamieson DJ, Schild L, Adams MM, Deshpande AD, Franks AL. Hospitalizations during pregnancy among managed care enrollees. Obstet Gynecol. 2002 Jul;100(1):94-100. doi: 10.1016/s0029-7844(02)02024-0. PMID 12100809
- [Background] Gadsby R, Barnie-Adshead AM, Jagger C. A prospective study of nausea and vomiting during pregnancy. Br J Gen Pract. 1993 Jun;43(371):245-8. PMID 8373648
- [Background] World Health Organisation, International Statistical Classification of Diseases and Related Health Problems. 10th Revision. Version for 2007.
- [Background] Nelson-Piercy C. Treatment of nausea and vomiting in pregnancy. When should it be treated and what can be safely taken? Drug Saf. 1998 Aug;19(2):155-64. doi: 10.2165/00002018-199819020-00006. PMID 9704251
- [Background] Goodwin TM, Montoro M, Mestman JH. Transient hyperthyroidism and hyperemesis gravidarum: clinical aspects. Am J Obstet Gynecol. 1992 Sep;167(3):648-52. doi: 10.1016/s0002-9378(11)91565-8. PMID 1382389
- [Background] Hod M, Orvieto R, Kaplan B, Friedman S, Ovadia J. Hyperemesis gravidarum. A review. J Reprod Med. 1994 Aug;39(8):605-12. PMID 7996524
- [Background] Bailit JL. Hyperemesis gravidarium: Epidemiologic findings from a large cohort. Am J Obstet Gynecol. 2005 Sep;193(3 Pt 1):811-4. doi: 10.1016/j.ajog.2005.02.132. PMID 16150279
- [Background] Ismail SK, Kenny L. Review on hyperemesis gravidarum. Best Pract Res Clin Gastroenterol. 2007;21(5):755-69. doi: 10.1016/j.bpg.2007.05.008. PMID 17889806
- [Background] Sheehan P. Hyperemesis gravidarum--assessment and management. Aust Fam Physician. 2007 Sep;36(9):698-701. PMID 17885701
- [Background] Verberg MF, Gillott DJ, Al-Fardan N, Grudzinskas JG. Hyperemesis gravidarum, a literature review. Hum Reprod Update. 2005 Sep-Oct;11(5):527-39. doi: 10.1093/humupd/dmi021. Epub 2005 Jul 8. PMID 16006438
- [Background] Oates-Whitehead R. Nausea and vomiting in early pregnancy. Clin Evid. 2004 Jun;(11):1840-52. No abstract available. PMID 15652084
- [Background] Alalade AO, Khan R, Dawlatly B. Day-case management of hyperemesis gravidarum: Feasibility and clinical efficacy. J Obstet Gynaecol. 2007 May;27(4):363-4. doi: 10.1080/01443610701327396. PMID 17654186
- [Background] Attkisson, C.C., and Greenfield, T. K. (1995). The Client Satisfaction Questionnaire (CSQ) scales and the Service Satisfaction Scale- 30 (SSS-30). In L.I. Sederer & B. Dickey (Eds.) Outcomes assessment in clinical practice. (pp. 120-127) Baltimore, MD: Williams & Wilkins. (SSS-30 is reproduced in Appendix pp. 279-283).
- [Background] Moher D, Schulz KF, Altman DG. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Lancet. 2001 Apr 14;357(9263):1191-4. PMID 11323066
- See also: Home page of Department of Obstetrics and Gynaecology, University College Cork, Cork University Maternity Hospital. — http://www.ucc.ie/en/obsgyn/